CLINICAL TRIAL: NCT06208189
Title: The Effect of Effort During a Resistance Exercise Session on Glycemic Control in Individuals With Prediabetes or Type 2 Diabetes Mellitus: a Randomized-controlled Trial
Brief Title: Is the Degree of Perceived Effort During Resistance Exercise Important for Improvements in Blood Glucose
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Flavio de Castro Magalhaes, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2310089095
Record Dates: First submitted 2023-12-28; First posted 2024-01-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes; Type 2 Diabetes Mellitus
Keywords: strength exercise; degree of effort; glycemic control; continuous glucose monitoring; prediabetes; type 2 diabetes mellitus
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized controlled, crossover, 3-way, clinical trial, following the SPIRIT and the TIDieR guidelines. After being considered eligible and agreeing to participate, participants will undergo anthropometrics assessment, familiarization sessions, and strength assessment before randomly carrying out 3 experimental (2 exercise and one control) periods, each composed of a total of ~48 hours, separated by at least 4 days. During the experimental periods diet will be strictly controlled and provided to the participants. Glycemic control will be assessed by a continuous glucose monitoring system throughout the experimental periods. The exercise sessions will be identical regarding total volume-load and session density, but proximity to failure in each set will be manipulated so effort will be different between the sessions. The control session will be identical in all procedures as the exercise sessions except that participants will remain sedentary.
Who Masked: Outcomes Assessor
Masking Description: Data and statistical analysis will be performed by a researcher blinded to groups and participants' identities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-effort session (Experimental): Participants will perform sets with as many repetitions they can each set.
  Interventions: Behavioral: High-effort session
- low-effort session (Experimental): Participants will perform sets with half of the anticipated number of repetitions of the high-effort session.
  Interventions: Behavioral: Low-effort session
- Control session (Sham Comparator): The control session all procedures will be identical to the high-effort session.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: High-effort session — Participants will perform 3 sets per exercise (total of 21 sets) with as many repetitions they can each set. We anticipate participants will perform ~10 repetitions per set in this session, with a total tempo of ~2.5 seconds per rep, averaging ~25 seconds per set. Resting period between exercises and sets will be 120 seconds. This will lead to a total session time of ~50 min. Their glycemic control will be evaluated during the following ~48 hours.
  Arms: high-effort session
Behavioral: Low-effort session — Participants will perform 6 sets per exercise (total of 42 sets) but perform half of the anticipated number of repetitions of the HIGH session (i.e., 5 reps). Repetition tempo at ~2.5 seconds will result in ~12.5 seconds per set. Resting period between exercises and sets will be 60 seconds. This prescription will also lead to a total session time of ~50 min. Thus, both the HIGH and LOW session will have similar total volume-load and session density, but differ in perceived effort after each set. Their glycemic control will be evaluated during the following ~48 hours.
  Arms: low-effort session
Behavioral: Control — The control session all procedures will be identical to the HIGH session, with the exception of performing the resistance exercises. However, to simulate all other procedures participants will follow all instructions, be positioned on the equipment for the same amount of time as the HIGH session, but will not perform any repetition. Interval between fake sets and exercises will be 120 seconds. Their glycemic control will be evaluated during the following ~48 hours.
  Arms: Control session

SUMMARY:
The goal of this clinical trial is to compare the degree of effort during a resistance exercise session on blood glucose levels in individuals with prediabetes or type 2 diabetes mellitus. The main questions it aims to answer are:

* Do individuals with prediabetes or type 2 diabetes mellitus need to perform resistance exercise with a high degree of effort for their blood glucose to improve?
* How do they feel (their enjoyment, discomfort) after the sessions with different degrees of effort?

Participants will perform 3 situations separated by at least 4 days, after being familiarized with all exercises and procedures:

* One control day, when they will not exercise;
* A high-effort resistance exercise session;
* A low-effort resistance exercise session Researchers will measure blood glucose levels and psychological responses after these situations to see if the effort was important for the improvement of their blood glucose and how effort affected the way they felt after each situation.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years;
* presence of prediabetes (fasting glycemia between 100 and 125 mg/dL or glycated hemoglobin [A1c] between 5.7 and 6.4%) or T2DM (fasting glycemia 126 mg/dL or above or A1c 6.5% or above).

Exclusion Criteria:

* renal failure,
* liver disease,
* uncontrolled hypertension (equal or greater than 160 mmHg systolic and/or equal or greater than 100 mmHg diastolic),
* history of severe cardiovascular problems,
* in case of oral hypoglycemic drugs usage, being on them for less than 6 months,
* inability to perform resistance exercise,
* being pregnant or trying to become pregnant during the course of the study,
* use of oral contraceptives,
* prisoners,
* persons requiring a legally authorized representative,
* non-English speakers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration | For 48 hours during each situation (arm) of the study
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)
Glucose concentration | For 6 hours during the morning (6 am - 12 pm) of each situation (arm) of the study
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)
Glucose concentration | For 6 hours during the afternoon (12 pm - 6 pm) of each situation (arm) of the study
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)
Glucose concentration | For 6 hours during the evening (6 pm - 12 am) of each situation (arm) of the study
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)
Glucose concentration | For 6 hours during the nocturnal period (12 am - 6 am) of each situation (arm) of the study
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)
Time in range | For 48 hours during each situation (arm) of the study
  Time of glucose concentration between 70 and 180 mg/dL (measured in minutes)
Time in range | For 6 hours during the morning (6 am - 12 pm) of each situation (arm) of the study
  Time of glucose concentration between 70 and 180 mg/dL (measured in minutes)
Time in range | For 6 hours during the afternoon (12 pm - 6 pm) of each situation (arm) of the study
  Time of glucose concentration between 70 and 180 mg/dL (measured in minutes)
Time in range | For 6 hours during the evening (6 pm - 12 am) of each situation (arm) of the study
  Time of glucose concentration between 70 and 180 mg/dL (measured in minutes)
Time in range | For 6 hours during the nocturnal period (12 am - 6 am) of each situation (arm) of the study
  Time of glucose concentration between 70 and 180 mg/dL (measured in minutes)
Prevalence of hyperglycemia | For 48 hours during each situation (arm) of the study
  Time of glucose concentrations >180 mg/dL (measured in minutes)
Prevalence of hyperglycemia | For 6 hours during the morning (6 am - 12 pm) of each situation (arm) of the study
  Time of glucose concentrations >180 mg/dL (measured in minutes)
Prevalence of hyperglycemia | For 6 hours during the afternoon (12 pm - 6 pm) of each situation (arm) of the study
  Time of glucose concentrations >180 mg/dL (measured in minutes)
Prevalence of hyperglycemia | For 6 hours during the evening (6 pm - 12 am) of each situation (arm) of the study
  Time of glucose concentrations >180 mg/dL (measured in minutes)
Prevalence of hyperglycemia | For 6 hours during the nocturnal period (12 am - 6 am) of each situation (arm) of the study
  Time of glucose concentrations >180 mg/dL (measured in minutes)
Prevalence of hypoglycemia | For 48 hours during each situation (arm) of the study
  Time of glucose concentrations <70 mg/dL (measured in minutes)
Prevalence of hypoglycemia | For 6 hours during the morning (6 am - 12 pm) of each situation (arm) of the study
  Time of glucose concentrations <70 mg/dL (measured in minutes)
Prevalence of hypoglycemia | For 6 hours during the afternoon (12 pm - 6 pm) of each situation (arm) of the study
  Time of glucose concentrations <70 mg/dL (measured in minutes)
Prevalence of hypoglycemia | For 6 hours during the evening (6 pm - 12 am) of each situation (arm) of the study
  Time of glucose concentrations <70 mg/dL (measured in minutes)
Prevalence of hypoglycemia | For 6 hours during the nocturnal period (12 am - 6 am) of each situation (arm) of the study
  Time of glucose concentrations <70 mg/dL (measured in minutes)

SECONDARY OUTCOMES:
Resistance Training Intensity by the Omni Perceived Exertion Scale | After each set of each exercise performed.
  Discrete scale from 0 to 10, where higher values mean more perceived exertion.
Feeling scale | Before and immediately after the resistance exercise sessions.
  Discrete scale from -5 to +5, where higher values mean more positive feelings.
Physical Activity Enjoyment Scale | Immediately after the resistance exercise sessions.
  Scale composed of 18 items, with scores from 1 to 7 each (total score from 18 to 126). After analysis, higher scores mean higher enjoyment.
Self-efficacy scale | Immediately after the resistance exercise sessions.
  Scale composed of 8 questions, with discrete options from 0 to 100%. Higher scores mean higher self-efficacy.
Rating of Discomfort scale | Before and 5 minutes after the resistance exercise sessions.
  Discrete scale from 0 to 100, where higher scores mean more discomfort.
Session rating of perceived exertion | 5 minutes after the resistance exercise sessions.
  Discrete scale from 0 to 10, where higher values mean more perceived exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio De Castro Magalhaes, PhD, Principal Investigator — Assistant Professor
Locations (1):
- UNM Exercise Physiology Lab, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
For sharing the data generated we will use the Open Science Framework (OSF) platform. Before data sharing, all personal identifiers will be stripped from the data. Specifically, any direct identifiers (e.g., name, email addresses, phone and cell phone numbers), date identifiers (e.g., birthday, date of disease diagnosis, dates patients participated in data collection), location identifiers (e.g., personal or professional addresses, zip codes), links to external datasets identifiers (e.g., social media accounts) will be removed. Furthermore, participants will be represented by an ID string generated randomly (https://www.random.org/strings/), and their data will be inserted in the files in a random order, not associated with the order they were enrolled. Thus, data will be entirely de-identified before sharing, in order to protect sensitive personal information and privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The anticipated date for data sharing will be 6 months after publication of data or 18 months after award end date, whatever happens first.
Access Criteria: Freely accesible.

REFERENCES:
- [Derived] Ramirez M, Gebauer M, Mermier C, Little JP, Lin L, Palley G, Hsiao YY, Mota Alvidrez RI, Mang ZA, Amorim FT, Tricoli V, De Castro Magalhaes F. The Effect of Effort During a Resistance Exercise Session on Glycemic Control in Individuals Living With Prediabetes or Type 2 Diabetes: Protocol for a Crossover Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 5;13:e63598. doi: 10.2196/63598. PMID 39499920